CLINICAL TRIAL: NCT05909501
Title: AGE-ING (Assessment of Geriatric Evaluations Impact on New AML Guidance) Study
Brief Title: Assessment of Geriatric Evaluations Impact on New AML Guidance
Acronym: AGE-ING
Status: Recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: UPCC 11423
Record Dates: First submitted 2023-06-12; First posted 2023-06-18 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: AML, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of the study is to measure physiologic age (there is no current formal definition but is meant to imply that patients should be evaluated holistically rather than on age alone) at baseline in newly diagnosed AML patients over 50 years receiving either intensive or non-intensive treatment. This information will be used to evaluate toxicity, early mortality, remission rates and long term survival.

ELIGIBILITY:
Inclusion Criteria:

* AML diagnosis by peripheral flow cytometry and/or bone marrow aspirate and biopsy
* New diagnosis being considered for new line of treatment
* Age ≥ 50 years.
* Performance status 0,1, and 2

Exclusion Criteria:

* Inability to understand or unable to sign a written informed consent
* Unable to fill out questionnaires on their own and/or do not have someone to help complete them

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the physician practices of Penn Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate physiologic age using baseline measures of physical function, depression, cognition, frailty, and PROs in newly diagnosed AML patients receiving intensive and non-intensive treatment in relation to overall survival at 1 year. | At baseline, 14 days after treatment, 1 month after treatment
  Short physical performance battery (SPPB), geriatric depression scale (GDS), mini-COG, patient reported outcomes of physical function, fatigue, depression, cognition, anxiety
Evaluate baseline measures of physiologic age in relation to short term mortality | At 30 days and 60 days
Evaluate baseline measures of physiologic age in relation to grade 3, 4, and 5 toxicities from treatment | At baseline, 14 days after treatment, 1 month after treatment
Evaluate baseline measures of physiologic age in relation to complete remission | At baseline, 14 days after treatment, 1 month after treatment
Compare baseline measurements to serial measurements to understand how physical function changes over time with treatment | At baseline, 14 days after treatment, 1 month after treatment
Evaluate albumin as a biomarker predictor of clinical outcomes of short term mortality, 1 year OS and toxicity | At 30 days and 60 days
Create a predictive pre-treatment screening tool | At baseline, 14 days after treatment, 1 month after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Lai, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center at University of Pennsylvania, Philadelphia, Pennsylvania, United States